CLINICAL TRIAL: NCT06565273
Title: Phase IIa Proof-of-Concept Study, With Dose-Titration Based on Treat-to-Target Strategy, to Investigate the Efficacy, Safety, and Tolerability of Subcutaneous Injection of Folate-based Liposomes Encapsulating Methotrexate (FBL-MTX) in Disease-modifying Antirheumatic Drugs (DMARD)-naïve Patients With Moderate-to-Severe Active Rheumatoid Arthritis and in Patients With an Inadequate Response or Intolerance to Oral MTX.
Brief Title: Study to Investigate the Efficacy, Safety, and Tolerability of FBL-MTX in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLFARCOS - Pharmaceutical and Cosmetic Solutions Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FBL-MTX-201
Record Dates: First submitted 2024-08-08; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FBL-MTX (Experimental): * DMARD-naïve Patients: Patients will be administered an initial dose of FBL-MTX of 1 mg, by SC route. Subsequent doses will be titrated according to clinical response at intervals of 4 weeks, for 12 weeks. Maximum dosage will be 2.5 mg, every 2 weeks.
  * Patients with an Inadequate Response or Intolerance to Oral MTX: Patients will be administered an initial dose of FBL-MTX 2.5 mg, by SC route. Subsequent doses will be titrated according to clinical response at intervals of 4 weeks, for 12 weeks. Maximum dosage will be 2.5 mg, every two weeks.
  Interventions: Drug: FBL-MTX

INTERVENTIONS:
Drug: FBL-MTX — Patients will be administered an initial dose of FBL-MTX by subcutaneous route. Subsequent doses will be titrated according to clinical response. Maximum dosage will be 2.5 mg, every 2 weeks.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of FBL-MTX administered by subcutaneous route in Rheumatoid Arthritis patients.

Participants will be screened within 28 days prior to treatment period, to confirm that they meet the selection criteria for the study.

Treatment period: The treatment period will consist of eight sequential study visits, separated by a 2-week interval.

* DMARD-naïve Patients: Patients will be administered an initial dose of FBL-MTX of 1 mg, by SC route. Subsequent doses will be titrated according to clinical response at intervals of 4 weeks, for 12 weeks. Maximum dosage will be 2.5 mg, every 2 weeks.
* Patients with an Inadequate Response or Intolerance to Oral MTX: Patients will be administered an initial dose of FBL-MTX 2.5 mg, by SC route. Subsequent doses will be titrated according to clinical response at intervals of 4 weeks, for 12 weeks. Maximum dosage will be 2.5 mg, every two weeks.

DETAILED DESCRIPTION:
The Sponsor is developing folate-based liposomes encapsulating methotrexate (FBL-MTX) as a putative therapy for RA, by intravenous (IV) or subcutaneous (SC) administration.

Considering the presented non-clinical and clinical data for FBL-MTX and that SC administration is the most adequate route for patient self-administration, the Sponsor intends to proceed the clinical development of FBL-MTX with the objective of providing a more patient-friendly product with at least the same efficacy.

This proof-of-concept study intends to demonstrate the plausibility of FBL-MTX SC administration in patients through the exploratory evaluation of SC FBL-MTX efficacy in patients with moderate-to-severe active RA, and collection data on its safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects with moderate-to-severe active RA, age ≥ 18 years, Body Mass Index > 35 kg/m2.
* Diagnosis of RA according to the 2010 classification criteria of the American College of Rheumatology/ European Alliance of Associations for Rheumatology, formerly known as European League Against Rheumatism, (ACR/EULAR), with a Total Score ≥ 6/10.
* At least moderately active disease, as defined by DAS28-CRP >3.2 at Screening and Baseline, including:
* Tender joint count (TJC) ≥ 4
* Swollen joint count (SJC) ≥ 4
* C Reactive protein (CRP) ≥ 5 mg/L
* Documented history of positive RA factor and/or cyclic citrullinated peptide antibody test.
* Chest X-ray performed in the previous 3 months not suggestive of tuberculosis.
* If under nonsteroidal anti-inflammatory drugs (NSAIDs), must be able to be on a stable regimen from at least 2 weeks before baseline up to end-of-study.
* If under an oral corticosteroid (≤ 10 mg per day of prednisone or equivalent), must be able to be on a stable regimen from at least 4 weeks before baseline up to EoS.
* Eligible to start treatment with an immunomodulator.
* No evidence of clinically significant active infection.

Exclusion Criteria:

* Positive Interferon-Gamma Release Assay (IGRA) test result.
* Creatinine clearance < 60 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Disease Activity Score (DAS) for 28-joint count using C-reactive protein (DAS28-CRP) at Week 14 | From screening up to week 14.
  The DAS28-CRP is a combined index for measuring disease activity in Rheumatoid Arthritis. The components of the DAS28-CRP assessment include: 28 tender and swollen joint counts, CRP, and Patient's Global Assessment of Disease Activity, using a visual analogue scale (VAS): DAS28-CRP = 0.56*sqrt(28*Tender Joint Count) + 0.28*sqrt(28*Swollen joint count) + 0.36*ln(C-Reactive protein+1) + 0.014* global visual analogue scale + 0.96; Note: The 28 joints examined and assessed as tender or not tender for TJC and as swollen or not swollen for SJC include 14 joints on each side of the participant's body: 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal joints, 2 interphalangeal joints of the thumb, 8 proximal interphalangeal joints, and 2 knees. Higher scores mean a worse outcome.
Change from baseline in DAS28-CRP at Weeks 4, 8, and 12. | From screening up to weeks 4, 8 and 12.
  The DAS28-CRP is a combined index for measuring disease activity in Rheumatoid Arthritis. The components of the DAS28-CRP assessment include: 28 tender and swollen joint counts, CRP, and Patient's Global Assessment of Disease Activity, using a visual analogue scale (VAS): DAS28-CRP = 0.56*sqrt(28*Tender Joint Count) + 0.28*sqrt(28*Swollen joint count) + 0.36*ln(C-Reactive protein+1) + 0.014* global visual analogue scale + 0.96; Note: The 28 joints examined and assessed as tender or not tender for TJC and as swollen or not swollen for SJC include 14 joints on each side of the participant's body: 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal joints, 2 interphalangeal joints of the thumb, 8 proximal interphalangeal joints, and 2 knees. Higher scores mean a worse outcome.
Number of subjects who achieve remission (DAS28-CRP <2.6) at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
  The DAS28-CRP is a combined index for measuring disease activity in Rheumatoid Arthritis. The components of the DAS28-CRP assessment include: 28 tender and swollen joint counts, CRP, and Patient's Global Assessment of Disease Activity, using a visual analogue scale (VAS): DAS28-CRP = 0.56*sqrt(28*Tender Joint Count) + 0.28*sqrt(28*Swollen joint count) + 0.36*ln(C-Reactive protein+1) + 0.014* global visual analogue scale + 0.96; Note: The 28 joints examined and assessed as tender or not tender for TJC and as swollen or not swollen for SJC include 14 joints on each side of the participant's body: 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal joints, 2 interphalangeal joints of the thumb, 8 proximal interphalangeal joints, and 2 knees. Higher scores mean a worse outcome.
Number of subjects who achieve low disease activity (DAS28-CRP <3.2) at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Number of subjects who achieve American College of Rheumatology (ACR) 20% (ACR20) response at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Number of subjects who achieve ACR50 response at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Number of subjects who achieve ACR70 response at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Change from baseline in Clinical Disease Activity Index (CDAI) at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Change from baseline in Simplified Disease Activity Index (SDAI) at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Change from baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) score at Weeks 4, 8, 12, and 14. | From screening up to weeks 4, 8, 12 and 14.
Change from baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) at Week 14. | From screening up to Week 14.

SECONDARY OUTCOMES:
Incidence of TEAEs and SAEs. Clinically relevant abnormalities in vital signs, 12-lead ECG, and laboratory parameters will be reported as AEs. | From date of screening until the date of the last post-study follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: José Costa, MD, Principal Investigator — Unidade Local de Saúde do Alto Minho, EPE
Locations (8):
- Portugal (8):
  - Unidade Local de Saúde da Região de Aveiro, EPE, Aveiro
  - Unidade Local de Saúde de Braga, EPE, Centro Clínico Académico de Braga (2CA-Braga), Braga
  - Unidade Local de Saúde da Guarda, EPE, Guarda
  - Unidade Local de Saúde do Alto Ave, EPE, Guimarães
  - Unidade Local de Saúde da Região de Leiria, EPE, Leiria
  - Unidade Local de Saúde do Alto Minho, EPE, Ponte de Lima
  - Unidade Local de Saúde de São João, EPE, Porto
  - Unidade Local de Saúde de Gaia e Espinho, EPE, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: No